CLINICAL TRIAL: NCT00264537
Title: A Multicenter, Randomized, Double-blind, Placebo-controlledTrial of Golimumab, a Fully Human Anti-TNFa MonoclonalAntibody, Administered Subcutaneously, in Methotrexate-naive Subjects With Active Rheumatoid Arthritis
Brief Title: A Study of the Safety and Efficacy of Golimumab in Subjects With Rheumatoid Arthritis That Are Methotrexate-naive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006331; GO-BEFORE; C0524T05
Record Dates: First submitted 2005-12-11; First posted 2005-12-13 (Estimated); Results first posted 2009-07-13 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Methotrexate Naïve; subcutaneous injection
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; golimumab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Placebo + Methotrexate (Experimental): Placebo subcutaneous injections (SC) every 4 weeks from Week 0 for up to 5 years (unless early escape at week 28); Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - if early escape, 50 mg SC injections every 4 weeks from Week 28 up to 5 years; Golimumab - Dr's discretion after unblinding (in participants receiving methotrexate plus placebo), 50 mg SC injections every 4 weeks up to 5 years; Golimumab- Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Placebo injections; Drug: Methotrexate capsules; Biological: Golimumab 50 mg injections; Biological: Golimumab 100 mg injections
- Group 2: Golimumab 100 mg + Placebo (Experimental): Golimumab 100 mg SC injections every 4 weeks from Week 0 for up to 5 years; placebo capsules weekly from Week 0 for up to 5 years (unless early escape at Week 28); Methotrexate - if early escape, 10 to 20 mg weekly from Week 28 up to 5 years; Methotrexate - Dr's discretion after unblinding (in participants receiving golimumab plus placebo) 10 to 20 mg weekly for up to 5 years; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Placebo capsules; Drug: Methotrexate capsules; Biological: Golimumab 50 mg injections; Biological: Golimumab 100 mg injections
- Group 3: Golimumab 50 mg + Methotrexate (Experimental): Golimumab 50 mg SC injections every 4 weeks from Week 0 for up to 5 years (unless early escape at week 28); Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - if early escape, 100 mg SC injections every 4 weeks from Week 28 for up to 5 yrs; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Methotrexate capsules; Biological: Golimumab 50 mg injections; Biological: Golimumab 100 mg injections
- Group 4: Golimumab 100 mg + Methotrexate (Experimental): Golimumab 100 mg SC injections every 4 weeks from Week 0 for up to 5 years; Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period will be until the week-52 database lock.
  Interventions: Drug: Methotrexate capsules; Biological: Golimumab 50 mg injections; Biological: Golimumab 100 mg injections

INTERVENTIONS:
Drug: Placebo injections — SC injections
  Arms: Group 1: Placebo + Methotrexate
Drug: Placebo capsules — Placebo capsules will be filled with microcrystalline cellulose (Avicel PH 102).
  Arms: Group 2: Golimumab 100 mg + Placebo
Drug: Methotrexate capsules — Methotrexate capsules will be filled with microcrystalline cellulose (Avicel PH 102) and a 2.5 mg methotrexate tablet.
Biological: Golimumab 50 mg injections — SC injections
Biological: Golimumab 100 mg injections — SC injections

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of golimumab, alone or in combination with methotrexate, as compared to methotrexate alone in rheumatoid arthritis subjects who have not been previously treated with methotrexate.

DETAILED DESCRIPTION:
Golimumab is a fully human protein (antibody) which binds to tumor necrosis factor (TNFa). TNFa is increased in patients with rheumatoid arthritis (RA), and plays a major role in causing the joint pain, swelling, and damage from RA. Other marketed drugs that target TNFa (anti-TNFa drugs) have been shown to be effective in reducing the symptoms, signs, and joint damage of RA, but have limitations with respect to safety and ease of use. This is a randomized, double-blind, placebo-controlled trial of the efficacy and safety of a new anti-TNFa drug, golimumab, at 2 doses, injected under the skin every 4 weeks, alone or in combination with methotrexate, compared with methotrexate alone, in subjects with active RA who have not been previously treated with methotrexate. The study hypothesis is that golimumab, alone or in combination with methotrexate, will be more effective in treatment of RA than methotrexate alone, as measured by the American College of Rheumatology (ACR) response criteria and change from baseline in van der Heide Modified Sharp (vdH-S) score, without causing unacceptable significant adverse effects. The ACR response criteria were designed to determine the percentage of subjects who have achieved a certain level of improvement in their signs and symptoms of rheumatoid arthritis. The vdH-S score is a measurement of the amount of joint damage in a subject as seen by x-ray. Other secondary measures of effectiveness include the Health Assessment Questionnaire (HAQ), which is a series of questions that measure a subject's impairment in physical function caused by RA. Golimumab 50 mg or 100 mg, or placebo injections under the skin every 4 weeks until Week52. Methotrexate (MTX) or placebo capsules will be given in addition. At Week52, subjects on MTX alone with joint pain or swelling get golimumab 50mg, and all subjects receive golimumab for about 4 more years.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) (according to the revised 1987 criteria of the ACR) for at least 3 months prior to first administration of study agent
* Are methotrexate (MTX)-naïve (ie, have not received more than 3 weekly doses of MTX for RA at any time)
* Have active RA as defined by persistent disease activity with at least 4 swollen and 4 tender joints, at the time of screening and baseline, and at least 2 of the following 4 criteria: a) C-reactive protein (CRP) >=1.5 mg/dL at screening or erythrocyte sedimentation rate (ESR) by Westergren method of >= 28 mm in the first hour at screening or baseline, b)Morning stiffness of >= 30 minutes at screening and baseline, c)Bone erosion by x-ray and/or MRI prior to first administration of study agent, d)Anti-cyclic citrullinated peptide (anti-CCP) antibody-positive or rheumatoid factor (RF) positive at screening
* If using oral corticosteroids, must be on a stable dose equivalent to <= 10 mg of prednisone/day for at least 2 weeks prior to first administration of study agent.

Exclusion Criteria:

* Can not have inflammatory diseases other than RA that might confound the evaluation of the benefit of golimumab therapy
* No treatment with disease-modifying anti-rheumatic drugs (DMARDs)/systemic immunosuppressives during the 4 weeks prior to the first administration of study agent
* No prior treatment with biologic anti-TNF drugs (infliximab, etanercept, adalimumab)
* No history of, or ongoing, chronic or recurrent infectious disease
* No serious infection within 2 months prior to first administration of study agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (75):
- United States (18):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Upland, California
  - Jacksonville, Florida
  - Miami, Florida
  - Coeur d'Alene, Idaho
  - Moline, Illinois
  - Springfield, Illinois
  - Kansas City, Kansas
  - Witchita, Kansas
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Charlotte, North Carolina
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - Fort Worth, Texas
  - Lubbock, Texas
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - Rosario
  - S.M. de Tucuman
  - San Miguel de Tucumán
- Australia (2):
  - Maroochydore
  - Melbourne
- Vienna, Austria
- Belgium (2):
  - Brussels
  - Liège
- Canada (2):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
- Chile (2):
  - Rancagua
  - Santiago
- Hungary (3):
  - Budapest
  - Gyula
  - Szombathely
- India (3):
  - Bangalore
  - Lucknow Gpo
  - Secunderabad
- Malaysia (3):
  - Precinct 7
  - Saemban
  - Selayang Baru Utara
- New Zealand (2):
  - Auckland
  - Timaru
- Philippines (3):
  - Cebu
  - Manila
  - Quezon
- Poland (5):
  - Bialystok
  - Elblag
  - Kalisz
  - Szczecin
  - Warsaw
- Russia (3):
  - Moscow
  - Saratov
  - Yaroslavl
- Singapore, Singapore
- South Korea (4):
  - Daejeon
  - Incheon
  - Seoul
  - Suwon
- Spain (4):
  - Madrid
  - Santander
  - Seville
  - Valencia
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Tiachung
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Ukraine (4):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kiev
- United Kingdom (2):
  - Leeds
  - London

REFERENCES:
- [Derived] Kay J, Fleischmann R, Keystone E, Hsia EC, Hsu B, Zhou Y, Goldstein N, Braun J. Five-year Safety Data from 5 Clinical Trials of Subcutaneous Golimumab in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, and Ankylosing Spondylitis. J Rheumatol. 2016 Dec;43(12):2120-2130. doi: 10.3899/jrheum.160420. Epub 2016 Nov 1. PMID 27803138
- [Derived] Baker JF, Conaghan PG, Emery P, Baker DG, Ostergaard M. Relationship of patient-reported outcomes with MRI measures in rheumatoid arthritis. Ann Rheum Dis. 2017 Mar;76(3):486-490. doi: 10.1136/annrheumdis-2016-209463. Epub 2016 Jul 18. PMID 27432355
- [Derived] Emery P, Fleischmann RM, Hsia EC, Xu S, Zhou Y, Baker D. Efficacy of golimumab plus methotrexate in methotrexate-naive patients with severe active rheumatoid arthritis. Clin Rheumatol. 2014 Sep;33(9):1239-46. doi: 10.1007/s10067-014-2731-y. Epub 2014 Jul 9. PMID 25005327
- [Derived] Emery P, Fleischmann RM, Doyle MK, Strusberg I, Durez P, Nash P, Amante E, Churchill M, Park W, Pons-Estel B, Xu W, Xu S, Wu Z, Hsia EC. Golimumab, a human anti-tumor necrosis factor monoclonal antibody, injected subcutaneously every 4 weeks in patients with active rheumatoid arthritis who had never taken methotrexate: 1-year and 2-year clinical, radiologic, and physical function findings of a phase III, multicenter, randomized, double-blind, placebo-controlled study. Arthritis Care Res (Hoboken). 2013 Nov;65(11):1732-42. doi: 10.1002/acr.22072. PMID 23861303
- [Derived] Ostergaard M, Emery P, Conaghan PG, Fleischmann R, Hsia EC, Xu W, Rahman MU. Significant improvement in synovitis, osteitis, and bone erosion following golimumab and methotrexate combination therapy as compared with methotrexate alone: a magnetic resonance imaging study of 318 methotrexate-naive rheumatoid arthritis patients. Arthritis Rheum. 2011 Dec;63(12):3712-22. doi: 10.1002/art.30592. PMID 22127693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 637 participants were enrolled at 90 centers: 25 sites in Asia, 34 sites in Europe/Australia/New Zealand, 10 sites in Latin America and 21 sites in North America.
Groups:
- Group 1: Placebo + Methotrexate: Placebo subcutaneous injections (SC) every 4 weeks from Week 0 for up to 5 years (unless early escape at week 28); Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - if early escape, 50 mg SC injections every 4 weeks from Week 28 up to 5 years; Golimumab - Dr's discretion after unblinding (in participants receiving methotrexate plus placebo), 50 mg SC injections every 4 weeks up to 5 years; Golimumab- Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
- Group 2: Golimumab 100 mg + Placebo: Golimumab 100 mg SC injections every 4 weeks from Week 0 for up to 5 years; placebo capsules weekly from Week 0 for up to 5 years (unless early escape at Week 28); Methotrexate - if early escape, 10 to 20 mg weekly from Week 28 up to 5 years; Methotrexate - Dr's discretion after unblinding (in participants receiving golimumab plus placebo) 10 to 20 mg weekly for up to 5 years; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
- Group 3: Golimumab 50 mg + Methotrexate: Golimumab 50 mg SC injections every 4 weeks from Week 0 for up to 5 years (unless early escape at week 28); Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - if early escape, 100 mg SC injections every 4 weeks from Week 28 for up to 5 yrs; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
- Group 4: Golimumab 100 mg + Methotrexate: Golimumab 100 mg SC injections every 4 weeks from Week 0 for up to 5 years; Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
Period: Overall Study
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate
Started | 160 | 159 | 159 | 159
Completed | 110 | 101 | 109 | 99
Not Completed | 50 | 58 | 50 | 60
Not completed — Death | 0 | 3 | 3 | 2
Not completed — Lost to Follow-up | 3 | 4 | 7 | 6
Not completed — Adverse Event | 21 | 32 | 24 | 34
Not completed — Unsatisfactory therapeutic effect | 5 | 6 | 5 | 7
Not completed — Other | 21 | 11 | 10 | 11
Not completed — Not treated | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Total
Number analyzed (Participants) | 160 | 159 | 159 | 159 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.91) | 48.2 (12.85) | 50.9 (11.32) | 50.2 (11.87) | 49.5 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 134 | 135 | 125 | 528
  Male | 26 | 25 | 24 | 34 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved American College of Rheumatology (ACR) 50 Response at Week 24
Description: ACR 50 response is defined as a greater than or equal to 50 percent improvement from baseline in: 1. Swollen joint count (66 joints) and tender joint count (68 joints) 2. greater than or equal to 50 percentage improvement in 3 of the following 5 assessments: a. Patient's assessment of pain by the Visual Analogue Scale (VAS) (0-10 cm) b.Patient's Global Assessment of Disease activity VAS (0-10 cm) c. Physician's Global Assessment of Disease Activity VAS (0-10 cm) d. Patient's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein.
Time Frame: Week 24
Population: All participants randomly assigned to each treatment group. Participants considered non-responders if used any prohibited medications or discontinued subcutaneous study agent due to lack of efficacy. Missing ACR components imputed by Last Observation Carried Forward unless all ACR components were missing; in which case considered non-responders.
Measure: Number; unit: Participants
Groups:
- Combined Golimumab + Methotrexate: Combines Group 3 (golimumab 50 mg + methotrexate) and Group 4 (golimumab 100 mg + methotrexate)
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 160 | 159 | 159 | 159 | 318
Participants | 47 | 52 | 64 | 58 | 122
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Null hypothesis: No difference in ACR 50 response comparing Group 1 vs combined Groups 3 and 4. The sample size of 150 patients per treatment group will provide >98% power to detect a difference in ACR 50 response between treatment groups at alpha=0.05, assuming 50% of patients with screening C-reactive protein (CRP)<1.5mg/dL, and the difference in ACR 50 response of 15-20% in patients with screening CRP<1.5mg/dL and 20-25% in subjects with screening CRP>=1.5mg/dL, between Groups 1 vs 3 or 4; Test type: Superiority or Other; p = 0.053, Cochran-Mantel-Haenszel — A positive test is concluded if there is a significant difference between golimumab+MTX and placebo+MTX and at least one of the pair-wise comparisons at a 0.05 level; Cochran-Mantel-Haenszel (CMH) test stratified by screening CRP (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Null hypothesis: No difference in ACR 50 response comparing Groups 1 vs 3; Test type: Superiority or Other; p = 0.042, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Null hypothesis: No difference in ACR 50 response comparing Groups 1 vs 4; Test type: Superiority or Other; p = 0.177, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Null hypothesis: Group 2 is inferior to Group 1. Noninferiority of golimumab will be demonstrated if the lower bound of the 2-sided 95% CI is above -10%. The 10% non-inferiority margin was chosen because this difference is not clinically admissible. Under the above noted assumed response rates, this corresponds to preservation of at least 70% [(33% - 10%)/33%*100] of the expected "MTX benefit"; Test type: Non-Inferiority or Equivalence — This sample size (150 patients per treatment group) will provide approximately 85% power to claim non-inferiority of golimumab alone (Group 2) compared with MTX alone (Group 1) at alpha= 0.05 using a one-sided equivalence test assuming the proportion of golimumab alone (Group 2) treated patients with ACR 50 response is not less than 10% compared with proportion of patients with ACR 50 response in MTX alone (Group 1) treated group; p = 0.521, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL); Difference in ACR 50 Response Rate(%) = 3.3, 95% CI [lower limit -6.8] (The upper bound of 95% CI was not produced because it was not relevant to the pre-specified analysis) — The positive difference indicates in favor of golimumab+placebo compared to placebo+MTX; The upper bound of CI is not applicable

2. Secondary Outcome: Number of Participants Who Achieved American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR 20 response is defined as a greater than or equal to 20 percent improvement from baseline in: 1. Swollen joint count (66 joints) and tender joint count (68 joints) 2. greater than or equal to 20 percentage improvement in 3 of the following 5 assessments: a. Patient's assessment of pain by the Visual Analogue Scale (VAS) (0-10 cm) b.Patient's Global Assessment of Disease activity VAS (0-10 cm) c. Physician's Global Assessment of Disease Activity VAS (0-10 cm) d. Patient's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 160 | 159 | 159 | 159 | 318
Participants | 79 | 82 | 98 | 98 | 196
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Test type: Superiority or Other; p = 0.011, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel(CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel; CMH test stratified by screening CRP (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel; CMH test stratified by screening CRP (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.677, Cochran-Mantel-Haenszel; CMH test stratified by screening CRP (< 1.5 mg/dL; >= 1.5 mg/dL)

3. Secondary Outcome: Number of Patients With Abnormal Baseline C-reactive Protein (CRP) Who Achieved American College of Rheumatology (ACR) 50 Response at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Randomized participants with abnormal baseline CRP. Participants considered non-responders if used any prohibited medications or discontinued subcutaneous study agent due to lack of efficacy. Missing ACR components imputed by Last Observation Carried Forward unless all ACR components were missing; in which case considered non-responders.
Measure: Number; unit: Participants
Groups:
- Group 4: Golimumab 100 mg + Methotrexate (MTX): Golimumab 100 mg SC injections every 4 weeks from Week 0 for up to 5 years; Methotrexate - 10 to 20 mg weekly from Week 0 for up to 5 years; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50mg. Duration of the blinded period was until the week-52 database lock.
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate (MTX) | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 95 | 90 | 86 | 83 | 169
Participants | 34 | 26 | 38 | 37 | 75
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Test type: Superiority or Other; p = 0.178, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p = 0.250, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate (MTX); Test type: Superiority or Other; p = 0.240, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel(CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.339, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel(CMH) test stratified by screening C-reactive protein (CRP) (< 1.5 mg/dL; >= 1.5 mg/dL)

4. Primary Outcome: Change From Baseline in Total Van Der Heijde Modified Sharp (vdH-S) Score at Week 52
Description: The vdH-S score is the sum of the joint erosion score and the joint-space narrowing (JSN) score. The total score ranges from 0 (best) to 448 (worst) with higher scores indicating more joint damage.
Time Frame: Baseline and Week 52
Population: All participants randomly assigned to each treatment group.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined Golimumab + Methotrexate
Number analyzed (Participants) | 160 | 159 | 159 | 159 | 318
Scores on a scale | 1.37 (4.555) | 1.25 (6.155) | 0.74 (5.233) | 0.07 (1.833) | 0.41 (3.929)
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined Golimumab + Methotrexate; Null Hypothesis: No difference in vdH-S score comparing Groups 1 vs Groups 3 and 4 combined. The sample size of 150 subjects in each treatment group (Group 1, Group 3, Group 4) will provide > 95% power to detect a difference in the vdH-S score between treatment groups using a 2-sided t-test on van der Waerden normal scores of change from baseline in vdH-S score at α = 0.05, assuming a mean change from baseline in vdH-S score of 3.5 for the placebo group and 1 for Groups 3 and 4; Test type: Superiority or Other; p = 0.006, ANOVA — If this test is significant, a pairwise comparison between Group 3 and Group 1, and between Group 4 and Group 1 will be performed; A 2-sided ANOVA on the van der Waerden normal scores with 1 factor: screening CRP (< 1.5 mg/dL; ≥ 1.5 mg/dL)
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Null hypothesis: No difference in vdH-S score comparing Groups 1 vs 3; Test type: Superiority or Other; p = 0.015, ANOVA; A 2-sided ANOVA on the van der Waerden normal scores with 1 factor: screening CRP (< 1.5 mg/dL; >= 1.5 mg/dL)
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Null hypothesis: No difference in vdH-S score comparing Groups 1 vs 4; Test type: Superiority or Other; p = 0.025, ANOVA; A 2-sided ANOVA on the van der Waerden normal scores with 1 factor: screening CRP (< 1.5 mg/dL; >= 1.5 mg/dL)

5. Secondary Outcome: Change From Baseline in Total Van Der Heijde Modified Sharp (vdH-S) Score at Week 52 in Patients With Abnormal C-reactive Protein (CRP Greater Than 1.0 mg/dL) at Baseline
Description: as for outcome 4
Time Frame: Baseline and Week 52
Population: All participants randomly assigned to each treatment group who had C-reactive protein > 1.0 mg/dl at baseline.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Combined: Golimumab + Methotrexate: Combines Group 3 (golimumab 50 mg + methotrexate) and Group 4 (golimumab 100 mg + methotrexate)
Arm/Group | Group 1: Placebo + Methotrexate | Group 2: Golimumab 100 mg + Placebo | Group 3: Golimumab 50 mg + Methotrexate | Group 4: Golimumab 100 mg + Methotrexate | Combined: Golimumab + Methotrexate
Number analyzed (Participants) | 160 | 159 | 159 | 159 | 318
Scores on a scale | 2.16 (5.642) | 2.19 (7.967) | 1.29 (6.991) | 0.16 (2.195) | 0.74 (5.235)
Statistical Analysis 1: Comparison: Group 1: Placebo + Methotrexate vs Combined: Golimumab + Methotrexate; Test type: Superiority or Other; p = 0.003, ANOVA; 2-sided ANOVA on the van der Waerden normal scores
Statistical Analysis 2: Comparison: Group 1: Placebo + Methotrexate vs Group 3: Golimumab 50 mg + Methotrexate; Test type: Superiority or Other; p = 0.010, ANOVA; 2-sided ANOVA on the van der Waerden normal scores
Statistical Analysis 3: Comparison: Group 1: Placebo + Methotrexate vs Group 4: Golimumab 100 mg + Methotrexate; Test type: Superiority or Other; p = 0.014, ANOVA; 2-sided ANOVA on the van der Waerden normal scores
Statistical Analysis 4: Comparison: Group 1: Placebo + Methotrexate vs Group 2: Golimumab 100 mg + Placebo; Test type: Superiority or Other; p = 0.545, ANOVA; 2-sided ANOVA on the van der Waerden normal scores

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 5 years
Description: 3 of 637 randomized participants did not receive treatment & additional 18 participants did not receive any treatment with golimumab during the study. Thus only 616 participants are included in 5-year safety data. AEs were planned to be reported in relation to the doses of golimumab received throughout the study, rather than the treatment regimen.
Groups:
- Group A: Golimumab 50 mg SC Injections Only: Participants who were treated with golimumab and received golimumab 50 mg injections only during the study. Participants also received methotrexate capsules throughout the study. Participants were included from Group 1 and Group 3, who received only Golimumab 50 mg SC Injections.
- Group B: Golimumab 100 mg SC Injections Only: Participants who were treated with golimumab and received golimumab 100 mg injections only during the study. Participants also received either methotrexate or placebo capsules throughout the study. Participants were included from Group 1, Group 2 and Group 4, who received only Golimumab 100 mg SC Injections.
- Group C: Golimumab 50 and 100 mg SC Injections: Participants who were treated with golimumab and received at least one injection of both golimumab 50 mg and golimumab 100 mg during the study. Participants also received either methotrexate or placebo capsules throughout the study. Participants were included from Group 1, Group 2, Group 3 and Group 4, who received Golimumab 50 mg and 100 mg SC Injections.
Arm/Group | Group A: Golimumab 50 mg SC Injections Only | Group B: Golimumab 100 mg SC Injections Only | Group C: Golimumab 50 and 100 mg SC Injections
Serious Adverse Events (participants affected / at risk) | 55/172 | 94/243 | 55/201
Other Adverse Events (participants affected / at risk) | 139/172 | 215/243 | 174/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Golimumab 50 mg SC Injections Only (N=172) | Group B: Golimumab 100 mg SC Injections Only (N=243) | Group C: Golimumab 50 and 100 mg SC Injections (N=201)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 2 | 1 | 0
Addison's Disease (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Retinal Artery Embolism (Eye disorders) | 0 | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 1 | 0
Injection Site Erythema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 1 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 3 | 1
Cholestasis of Pregnancy (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 1 | 1 | 2
Arthritis Bacterial (Infections and infestations) | 0 | 1 | 0
Bone Tuberculosis (Infections and infestations) | 1 | 0 | 0
Breast Abscess (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Bursitis Infective (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Dengue Fever (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Encephalitis Viral (Infections and infestations) | 0 | 1 | 0
Enteritis Infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
H1n1 Influenza (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 2 | 3
Intervertebral Discitis (Infections and infestations) | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 2 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 1
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 1 | 0
Peritoneal Tuberculosis (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis JiroveCI Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 4 | 5
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 4 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 3 | 1
Septic Shock (Infections and infestations) | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 2 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 1
Tuberculosis Gastrointestinal (Infections and infestations) | 0 | 2 | 0
Tuberculous Pleurisy (Infections and infestations) | 0 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 2
Vulval Abscess (Infections and infestations) | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Face Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Open Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Synovial Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
General Physical Condition Abnormal (Investigations) | 0 | 1 | 0
Weight Increased (Investigations) | 0 | 0 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 6 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 2 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Demyelination (Nervous system disorders) | 0 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Multiple Sclerosis (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 4 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0 | 0
Bipolar I Disorder (Psychiatric disorders) | 1 | 0 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0
Delusional Disorder, Unspecified Type (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Bladder Prolapse (Renal and urinary disorders) | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urethral Disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Breast Calcifications (Reproductive system and breast disorders) | 0 | 1 | 0
Breast Inflammation (Reproductive system and breast disorders) | 0 | 0 | 1
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine Cervical Squamous Metaplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alveolitis Fibrosing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epiglottic Cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rheumatoid Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Generalised Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arterial Stenosis (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Femoral Arterial Stenosis (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Iliac Artery Stenosis (Vascular disorders) | 0 | 1 | 0
Varicose Ulceration (Vascular disorders) | 0 | 0 | 1
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Golimumab 50 mg SC Injections Only (N=172) | Group B: Golimumab 100 mg SC Injections Only (N=243) | Group C: Golimumab 50 and 100 mg SC Injections (N=201)
Anaemia (Blood and lymphatic system disorders) | 5 | 9 | 11
Abdominal Pain (Gastrointestinal disorders) | 10 | 11 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 20 | 17
Diarrhoea (Gastrointestinal disorders) | 15 | 17 | 17
Dyspepsia (Gastrointestinal disorders) | 18 | 17 | 21
Gastritis (Gastrointestinal disorders) | 7 | 16 | 10
Nausea (Gastrointestinal disorders) | 22 | 55 | 44
Vomiting (Gastrointestinal disorders) | 8 | 17 | 18
Fatigue (General disorders) | 7 | 21 | 10
Injection Site Erythema (General disorders) | 10 | 28 | 12
Pyrexia (General disorders) | 4 | 13 | 14
Bronchitis (Infections and infestations) | 26 | 40 | 34
Gastroenteritis (Infections and infestations) | 9 | 11 | 13
Influenza (Infections and infestations) | 12 | 17 | 16
Nasopharyngitis (Infections and infestations) | 20 | 31 | 33
Oral Herpes (Infections and infestations) | 7 | 2 | 12
Pharyngitis (Infections and infestations) | 16 | 27 | 20
Respiratory Tract Infection (Infections and infestations) | 9 | 11 | 5
Sinusitis (Infections and infestations) | 26 | 19 | 24
Upper Respiratory Tract Infection (Infections and infestations) | 45 | 62 | 72
Urinary Tract Infection (Infections and infestations) | 15 | 28 | 16
Alanine Aminotransferase Increased (Investigations) | 31 | 36 | 32
Aspartate Aminotransferase Increased (Investigations) | 21 | 21 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 21 | 17
Back Pain (Musculoskeletal and connective tissue disorders) | 17 | 23 | 22
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 19 | 11
Dizziness (Nervous system disorders) | 6 | 15 | 8
Headache (Nervous system disorders) | 14 | 33 | 16
Paraesthesia (Nervous system disorders) | 4 | 7 | 11
Depression (Psychiatric disorders) | 16 | 10 | 21
Insomnia (Psychiatric disorders) | 4 | 17 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 37 | 29
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 12 | 14
Rash (Skin and subcutaneous tissue disorders) | 9 | 18 | 15
Hypertension (Vascular disorders) | 19 | 25 | 23

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in less than or equal to 5% of patients. This information may vary from existing approved labeling and publications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.